CLINICAL TRIAL: NCT07034469
Title: Gas Tamponade Versus Air During Vitrectomy for Rhegmatogenous rEtinal dEtachmeNt; a Randomised Controlled Trial
Brief Title: Air Tamponade Versus Fluorinated Gas Tamponade for Rhegmatogenous Retinal Detachment
Acronym: GREEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHS0250
Record Dates: First submitted 2024-12-19; First posted 2025-06-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Retinal Detachment Rhegmatogenous
Keywords: retinal detachment; gas tamponade; air
MeSH Terms: conditions — Retinal Detachment | interventions — Air; Sulfur Hexafluoride

STUDY DESIGN:
Intervention Model Description: one arm will have standard of care gas tamponade, the study arm will have air tamponade
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterile air tamponade (Experimental): use of sterile air in place of fluorinated gases as a tamponade agent for rhegmatogenous retinal detachment vitrectomy surgery
  Interventions: Procedure: air
- Fluorinated gas tamponade (Active Comparator): use of fluorinated gas (SF6, C2F6 or C3F8) as a tamponade agent for rhegmatogenous retinal detachment treated with vitrectomy
  Interventions: Procedure: Gas SF6 (Sulfur Hexafluoride) and others

INTERVENTIONS:
Procedure: air — use of sterile air as a tamponade
  Arms: Sterile air tamponade
Procedure: Gas SF6 (Sulfur Hexafluoride) and others — use of fluorinated gases such as SF6, C2F6 or C3F8 as a tamponade agent
  Arms: Fluorinated gas tamponade

SUMMARY:
TITLE: RCT of air tamponade versus fluorinated gas tamponade for rhegmatogenous retinal detachment DESIGN: Non-inferiority RCT of 150 patients from 10 UK centres AIMS: To assess whether air tamponade is non inferior to gas tamponade for the repair of RRD treated with vitrectomy.

PRIMARY OUTCOME MEASURE: Primary anatomical success with single operation at 24 weeks.

DETAILED DESCRIPTION:
STUDY OBJECTIVES To assess whether air tamponade is non inferior to gas tamponade for the repair of RRD with superior breaks treated with vitrectomy and to assess how cost-effective air tamponade is compared to gas tamponade BACKGROUND Rhegmatogenous retinal detachment (RRD) is the most common form of RD developing when there is a retinal 'break' that allows the ingress of fluid from the vitreous cavity into the subretinal space. There are three main current options for the management of RRD, namely pneumoretinopexy, scleral buckling and vitrectomy (PPV). Vitrectomy is currently performed for the majority of RRDs in the UK. Tamponade in PPV is usually performed by complete filling of the vitreous cavity with fluorinated gases diluted in air at iso-volumetric concentrations which do not expand (e.g., 20% SF6 or 14% C3F8).

RATIONALE FOR CURRENT STUDY The use of air instead of fluorinated gases in primary RRD treated with vitrectomy has been the subject of much debate recently. Air being non expansile and short lived it offers the prospect of quicker rehabilitation and less risk and avoids the use of environmentally damaging fluorinated gases. The question of whether air offers equivalence to gas for uncomplicated RRD with mainly superior breaks has not been adequately answered, as reviewed in a recent systematic review and meta-analysis where the certainty of evidence was judged very low. This type of detachment is the commonest at approximately 60% of the cases in the BEAVRS database and representing approximately 4,800 RRD in the UK per annum. There has been significant interest in air recently with the announcement of the European chemical agencies proposed ban on fluorinated gases.

There are several potential benefits of using air over gas to repair detached retinas.

1. Speedier visual recovery, which may mean earlier return to work or normal activities.
2. Avoiding expansile fluorinated gas-related complications such as raised eye pressure, reducing the number of post-operative visits and medications needed after surgery.
3. Fewer restrictions after surgery (able to fly and drive sooner and shorter restrictions on anaesthetic agents)
4. Decreased environmental impact by reducing greenhouse gas use. If air was proven to be non-inferior to gas, then patients with RRD treated by vitrectomy would likely prefer it STUDY DESIGN RCT of people presenting with uncomplicated RRD treated with vitrectomy comparing air to gas tamponade.

Participants will be randomised 1:1 between air tamponade and gas tamponade. Randomisation will be performed using a secure web-based randomisation system at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary uncomplicated RRD undergoing vitrectomy.
* Phakic and pseudophakic eyes
* Retinal breaks superiorly between 3 and 9 o'clock, and that are separated by less than 4 clock hours.

Exclusion Criteria:

* Absence of PVD
* Age 40 years or younger
* PVR grade C or above
* Aphakia or anterior chamber lens
* Retinal breaks greater than 1 clock hour in size
* Retinal breaks that exist below 3 and 9 o'clock on both the nasal and temporal sides.
* Retinal breaks at or posterior to the vessel arcades
* Current or previous -6D myopia or greater (or axial length >26millimetres (mm))
* Chronic RRD judged by the presence of subretinal bands and other signs of -chronicity or by history of visual loss for >28 days.
* Significant inflammation, choroidal detachments, hypotony (<6 millimetres of mercury (mmHg) preop)
* Previous open-globe injury, or endophthalmitis
* Current or previous posterior uveitis or choroiditis
* Any intraocular surgical procedure within 4 weeks other than laser/cryotherapy
* Any other condition that, in the opinion of the investigator, would prevent the participant from granting informed consent or complying with the protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2029-03-20 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Primary anatomical success | 6 months
  Primary anatomical success at 24 weeks assessed by clinical examination by a retinal surgeon. The Outcome is binary with either 'successful retinal reattachement' or 'failed surgery'

SECONDARY OUTCOMES:
Post op visual acuity | 10 days, 6 weeks and 24 weeks
  Postoperative visual acuity at 10 days, 6 and 24 weeks measured either in Snellen or logMAR
Intraocular pressure | Day 1, 10 and 6 and 24 weeks
  Day 1, Day 10-, 6- and 24-weeks intraocular pressure measured in mmHg
Quality of Life measures | 10 days, 6 and 24 weeks
  Generic and vision related quality of life using the Euro quality of Life and Visual function questionnaire at 10 days, 6 and 24 weeks postoperatively. These questionnaires have sections relating to ocular health eg vision, ocular pain etc and impact on daily activities. They create a composite score combining each section, which ranges from 0-100 with higher scores reflecting better vision related quality of life.
Patient Satisfaction | 10 days, 6 and 24 weeks
  Patient satisfaction with treatment using the Macular Disease Treatment Satisfaction Questionnaire at 10 days, 6 and 24 weeks. This questionnaire is a self administered questionnaire with a 7 point (0-6) scoring over 14 domains with a total score of 0-72, with higher scores reflecting greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Rumana N Hussain, MBBS, FRCOph, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust UK

IPD SHARING:
Plan to Share IPD: No